CLINICAL TRIAL: NCT01877148
Title: Effects of Transcranial Direct Current Stimulation Associated With Physical Therapy on Motor Rehabilitation in Parkinson´s Disease Patients
Brief Title: Effects Of tDCS With Physical Therapy On Rehabilitation In Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Doctor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Parkinson_tDCS_rehabilitation
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2013-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson, rehabilitation, tDCS
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiotherapy + anodal tDCS (Experimental): The patients will be submit to anodal tDCS applied in the motor cortex and after the patient will be submit to a 30 minutes of physiotherapy protocol.
  Interventions: Device: tDCS; Behavioral: Physiotherapy
- Physiotherapy + sham tDCS (Sham Comparator): The patients will be submit to sham tDCS and after the patient will be submit to a 30 minutes of physiotherapy protocol.
  Interventions: Device: tDCS; Behavioral: Physiotherapy

INTERVENTIONS:
Device: tDCS — tDCS involves application of very low amplitude direct current via surface scalp electrodes. The applied current modifies the transmembrane neuronal potential and thus influences the level of excitability. Depending on the polarity of active electrodes tDCS can increase or decrease the cortical excitability. The anodal tDCS increase the excitability.
  Other Names: non invasive brain stimulation
Behavioral: Physiotherapy — Physiotherapy protocol followed the guidelines outlined in clinical practice guideline for physical therapy in Parkinson disease of the Royal Dutch society for physical therapy (Keus, 2007). This guideline proposes some objectives for motor rehabilitation in patients with PD, such as: flexibility, strength, coordination, balance, posture and gait. The difficulty of exercises ranged according with Hoehn and Yahr (HY) staging scale. In this way, each stage of HY had a specific physical therapy protocol following the guideline.

SUMMARY:
The present study aims to investigate the effect of transcranial direct current stimulation (tDCS) associated with physiotherapy in parkinson´s rehabilitation. Previous studies showed that tDCS could reduce the bradykinesia, one of the symptom of Parkinson disease. In this way, this study will combine tDCS with physiotherapy in order to enhance the motor rehabilitation and the quality of life.

DETAILED DESCRIPTION:
12 patients were participated of this study.After screening to check the eligibility criteria and giving informed consent, they were randomized in two groups. All patients were submitted to a 10 therapeutic sessions that occurred 3 times per week.

Before, immediately after and 1 month after the last session patients were submitted to an evaluation with the follow tests: Unified Parkinson´s Disease Rating Scale(UPDRS), Jebsen Taylor Test (JTT) and Parkinson's Disease Quality of Life (PDQL). Furthermore, before and after each session the patients were submitted to transcranial magnetic stimulation (TMS) to evaluate cortical excitability through motor threshold and motor evoked potential.

In experimental sessions, the subjects always received physiotherapy with conventional techniques, the protocol followed the clinical practice guideline for physical therapy in Parkinson disease with the Royal Dutch Society Therapy. During tDCS protocol the patients seated in a comfortable chair with head and arm rests. Continuous current was applied using a pair of saline-soaked surface sponge electrodes (surface 35 cm2), the anode electrode was placed over the primary motor cortex and cathode above contralateral orbit. tDCS was applied of twice stimulation of 13 minutes with 20 minutes of interval between them and a current strength of 1mA. Sham tDCS was applied by current flow of 30s.

ELIGIBILITY:
Inclusion Criteria:

Parkinson disease comproved by a neurologist Regular treatment with dopamine or other drugs against parkinson -

Exclusion Criteria:

pregnant history of convulsion metal implant in the region of skull or face change in medication during the study realize other physical therapy in the same time of the study previous surgery for parkinson disease

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kátia K Monte-Silva, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Physiotherapy + Anodal tDCS: The patients will be submit to anodal tDCS applied in the motor cortex and after the patient will be submit to a 30 minutes of physiotherapy protocol.
  Transcranial direct current stimulation: tDCS involves application of very low amplitude direct current via surface scalp electrodes. The applied current modifies the transmembrane neuronal potential and thus influences the level of excitability. Depending on the polarity of active electrodes tDCS can increase or decrease the cortical excitability. The anodal tDCS increase the excitability
  Physiotherapy
- Physiotherapy + Sham tDCS: The patients will be submit to sham tDCS and after the patient will be submit to a 30 minutes of physiotherapy protocol.
  Transcranial direct current stimulation: tDCS involves application of very low amplitude direct current via surface scalp electrodes. The applied current modifies the transmembrane neuronal potential and thus influences the level of excitability. Depending on the polarity of active electrodes tDCS can increase or decrease the cortical excitability. The anodal tDCS increase the excitability
  Physiotherapy
Period: Overall Study
Arm/Group | Physiotherapy + Anodal tDCS | Physiotherapy + Sham tDCS
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physiotherapy + Anodal tDCS | Physiotherapy + Sham tDCS | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9.27) | 68.2 (11.75) | 63.6 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  Brazil | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Unified Parkinson´s Disease Rating Scale - UPDRS
Description: Unified Parkinson´s Disease Rating Scale is the sum of 27 questions, total score ranging from108 (best possible outcome) to 0 (worst possible outcome)", as accurate and appropriate
Time Frame: At baseline, after 1 month
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Physiotherapy + Anodal tDCS | Physiotherapy + Sham tDCS
Number analyzed (Participants) | 5 | 5
units on a scale
  Baseline | 24 (12) | 30 (23)
  post 1 month | 21.2 (11.12) | 21.8 (14.0)

2. Secondary Outcome: Change From Cortical Excitability Via Single Transcranial Magnetic Stimulation
Time Frame: per sesssion: at baseline and after physical therapy
Measure: Mean (Standard Error); unit: milivolt
Arm/Group | Physiotherapy + Anodal tDCS | Physiotherapy + Sham tDCS
Number analyzed (Participants) | 5 | 5
milivolt
  Baseline | 1.01 (0.25) | 1 (0.22)
  post 1 month | 1.35 (0.24) | 1.15 (0.31)

3. Other Pre Specified Outcome: Change From Parkinson Disease Quality of Life - PDQL
Description: Parkinson disease quality of life is the sum of 37 questions, total score ranging from 0 (best possible outcome) to 185 (worst possible outcome)", as accurate and appropriate
Time Frame: at baseline, after 1 month
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Physiotherapy + Anodal tDCS | Physiotherapy + Sham tDCS
Number analyzed (Participants) | 5 | 5
units on a scale
  Baseline | 112.8 (44.1) | 117.2 (45.6)
  post 1 month | 120.2 (35.07) | 125.8 (37.83)

4. Other Pre Specified Outcome: Change From Jebsen-Taylor Hand Function Test - Jebsen Test
Description: The Jebsen-Taylor Hand Function Test assesses a broad range of uni-manual hand functions required for activities of daily living. Seven subtests are performed on both non-dominant and dominant hand: 1. Writing a 24-letter, 3rd grade reading difficulty sentence 2... Total score = sum of times for each subtests. Shorted times are indicative of better hand function
Time Frame: At baseline, after 1 month
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Physiotherapy + Anodal tDCS | Physiotherapy + Sham tDCS
Number analyzed (Participants) | 5 | 5
minutes
  Baseline | 106.36 (55.93) | 90.63 (45.53)
  post 1 month | 86.62 (48.71) | 81.29 (27.5)

ADVERSE EVENTS:
Time Frame: after tDCS
Description: Questionnaire of adverses effects
Arm/Group | Physiotherapy + Anodal tDCS | Physiotherapy + Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No